CLINICAL TRIAL: NCT04446273
Title: Effects of Proximal Priority Versus Distal Priority Robotic Priming Technique With Rehabilitation Therapy of Upper-Limb Functions in Patients With Chronic Stroke
Brief Title: Proximal Priority Versus Distal Priority Robotic Priming Effects in Patients With Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202004105RINB
Record Dates: First submitted 2020-06-18; First posted 2020-06-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Upper extremity rehabilitation; Proximal priority; Distal priority; Robotic therapy; Bilateral motor priming; Impairment-oriented training; Task-oriented training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into the proximal priority robotic priming and impairment-oriented training or the distal priority robotic priming and impairment-oriented training groups and receive 18 intervention sessions
Who Masked: Outcomes Assessor
Masking Description: Initial and outcome assessments will be administered by a well-trained and certified occupational therapist who is blinded to the group assignment, study hypotheses, and intervention of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRI group (Experimental): The PRI and DRI groups will receive an equal amount of treatment time, comprising 1.5 hours per day, 3 days per week, for 6 weeks. The PRI protocol provides robotic training for 45 minutes and impairment-oriented training for 45 minutes. The PRI group will start from the Bi-Manu-Track proximal mode (i.e., forearm) and then the Bi-Manu-Track distal mode (i.e., wrist).
  Interventions: Device: Bi-Manu-Track
- DRI group (Active Comparator): The PRI and DRI groups will receive an equal amount of treatment time, comprising 1.5 hours per day, 3 days per week, for 6 weeks. The DRI protocol provides robotic training for 45 minutes and impairment-oriented training for 45 minutes. The DRI group will start from the Bi-Manu-Track distal mode (i.e., wrist) and then the Bi-Manu-Track proximal mode (i.e., forearm).
  Interventions: Device: Bi-Manu-Track

INTERVENTIONS:
Device: Bi-Manu-Track — The PRI and DRI protocol provide robotic training for 45 minutes and impairment-oriented training for 45 minutes. The PRI group will start from the Bi-Manu-Track proximal mode (i.e., forearm) and then the Bi-Manu-Track distal mode (i.e., wrist). The DRI group will start from the Bi-Manu-Track distal mode (i.e., wrist) and then the Bi-Manu-Track proximal mode (i.e., forearm).In every session of robotic training, the patient will practice bilateral passive range of motion exercise, in which affected upper extremity is assisted by the unaffected side, and bilateral active range of motion exercise. Robotic training will be followed by impairment-oriented training.
  Other Names: impairment-oriented training

SUMMARY:
This is a single-blind randomized comparative efficacy study involving 54-72 participants with chronic stroke. Participants will be randomized into proximal priority robotic group or distal priority robotic group and receive 18 intervention sessions (90 min/d, 3 d/wk for 6 weeks). The Fugl-Meyer Assessment Upper Extremity subscale, Medical Research Council Scale, Revised Nottingham Sensory Assessment, and Wolf Motor Function Test will be administered at baseline, after treatment, and at the 3-month follow-up. Two-way repeated-measures analysis of variance and the Chi-Square Automatic Interaction Detector Method will be used to examine the comparative efficacy and predictors of outcome, respectively, after intervention.

DETAILED DESCRIPTION:
Background. The sequence of establishing proximal stability or function before facilitation of the distal body part has long been recognized in stroke rehabilitation practice but lacks scientific evidence. This study plans to examine the effects of proximal priority robotic priming and impairment-oriented training (PRI) and distal priority robotic priming and impairment-oriented training (DRI).

Methods. This is a single-blind randomized comparative efficacy study involving 54-72 participants with chronic stroke. Participants will be randomized into PRI or DRI groups and receive 18 intervention sessions (90 min/d, 3 d/wk for 6 weeks). The Fugl-Meyer Assessment Upper Extremity subscale, Medical Research Council Scale, Revised Nottingham Sensory Assessment, and Wolf Motor Function Test will be administered at baseline, after treatment, and at the 3-month follow-up. Two-way repeated-measures analysis of variance and the Chi-Square Automatic Interaction Detector Method will be used to examine the comparative efficacy and predictors of outcome, respectively, after PRI and DRI.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are age between 20 and 75 years old, more than 3 months after the onset of a first unilateral ischemic or hemorrhagic stroke, moderate to severe UE motor impairment (i.e., total UE score of the Fugl-Meyer Assessment [FMA] score between 18 and 56), no severe spasticity in any joints of the affected arm (modified Ashworth Scale score <3 in any of the affected shoulder, elbow, wrist, and fingers), able to follow instructions (Mini-Mental State Examination total score >24), no UE fractures in the past 3 months, and not simultaneously participating in other medication or rehabilitation studies.

Exclusion Criteria:

* The exclusion criteria are other neurologic, neuromuscular, or orthopedic disease, such as epilepsy, or severe health or physical conditions that might impede participation in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Fugl-Meyer Assessment will be administered to participants at baseline.
  Fugl-Meyer Assessment is used to assess motor impairment of body function, including ranges of motion of the upper extremity (UE) joints, and grasping, coordination, and speed of UE. movement.
Fugl-Meyer Assessment | Fugl-Meyer Assessment will be administered to participants at immediately after intervention.
  Fugl-Meyer Assessment is used to assess motor impairment of body function, including ranges of motion of the UE joints, and grasping, coordination, and speed of UE movement.
Fugl-Meyer Assessment | Fugl-Meyer Assessment will be administered to participants at three months after intervention.
  Fugl-Meyer Assessment is used to assess motor impairment of body function, including ranges of motion of the UE joints, and grasping, coordination, and speed of UE. movement.
Medical Research Council Scale | Medical Research Council Scale will be administered to participants at baseline.
  Medical Research Council Scale is used to assess muscle power of the affected upper extremity joints.
Medical Research Council Scale | Medical Research Council Scale will be administered to participants immediately after intervention.
  Medical Research Council Scale is used to assess muscle power of the affected upper extremity joints.
Medical Research Council Scale | Medical Research Council Scale will be administered to participants three months after intervention.
  Medical Research Council Scale is used to assess muscle power of the affected upper extremity joints.

SECONDARY OUTCOMES:
The ABILHAND Questionnaire | The ABILHAND Questionnaire will be administered to participants at baseline.
  The ABILHAND Questionnaire is an inventory of 23 manual activities on which the patient provides his or her self-perceived performing difficulty on a 3-level scale (impossible, difficult, easy).
The ABILHAND Questionnaire | The ABILHAND Questionnaire will be administered to participants immediately after intervention..
  The ABILHAND Questionnaire is an inventory of 23 manual activities on which the patient provides his or her self-perceived performing difficulty on a 3-level scale (impossible, difficult, easy).
The ABILHAND Questionnaire | The ABILHAND Questionnaire will be administered to participants three months after intervention..
  The ABILHAND Questionnaire is an inventory of 23 manual activities on which the patient provides his or her self-perceived performing difficulty on a 3-level scale (impossible, difficult, easy).
The Stoke Impact Scale 3.0 | The Stoke Impact Scale 3.0 will be administered to participants at baseline.
  The Stoke Impact Scale 3.0 is a 59-item questionnaire that measures perceived disability and health-related quality of life after stroke in eight domains: strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion, memory/thinking, and participation/role function.
The Stoke Impact Scale 3.0 | The Stoke Impact Scale 3.0 will be administered to participants immediately after intervention.
  The Stoke Impact Scale 3.0 is a 59-item questionnaire that measures perceived disability and health-related quality of life after stroke in eight domains: strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion, memory/thinking, and participation/role function.
The Stoke Impact Scale 3.0 | The Stoke Impact Scale 3.0 will be administered to participants three months after intervention.
  The Stoke Impact Scale 3.0 is a 59-item questionnaire that measures perceived disability and health-related quality of life after stroke in eight domains: strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion, memory/thinking, and participation/role function.
The Stroke Self-Efficacy Questionnaire | The Stroke Self-Efficacy Questionnaire will be administered to participants at baseline.
  The Stroke Self-Efficacy Questionnaire is a 13-item questionnaire to evaluate self-efficacy in functioning after stroke.
The Stroke Self-Efficacy Questionnaire | The Stroke Self-Efficacy Questionnaire will be administered to participants immediately after intervention.
  The Stroke Self-Efficacy Questionnaire is a 13-item questionnaire to evaluate self-efficacy in functioning after stroke.
The Stroke Self-Efficacy Questionnaire | The Stroke Self-Efficacy Questionnaire will be administered to participants three months after intervention.
  The Stroke Self-Efficacy Questionnaire is a 13-item questionnaire to evaluate self-efficacy in functioning after stroke.
The Wolf Motor Function Test | The Wolf Motor Function Test will be administered to participants at baseline.
  The Wolf Motor Function Test is used to assess functional motor ability of the upper extremity with 15 functional tasks.
The Wolf Motor Function Test | The Wolf Motor Function Test will be administered to participants immediately after intervention.
  The Wolf Motor Function Test is used to assess functional motor ability of the upper extremity with 15 functional tasks.
The Wolf Motor Function Test | The Wolf Motor Function Test will be administered to participants three months after intervention.
  The Wolf Motor Function Test is used to assess functional motor ability of the upper extremity with 15 functional tasks.
The Montreal Cognitive Assessment | The Montreal Cognitive Assessment will be administered to participants at baseline.
  The Montreal Cognitive Assessment is a cognitive screening assessment that is used to measure several cognitive domains, which include working memory, delayed recall, visuospatial abilities, executive functions, attention, concentration, language, and orientation to time and place. The total score ranges from 0 to 30. One extra point is added to adjust the total score for participants who received less than 12 years of education.
The Montreal Cognitive Assessment | The Montreal Cognitive Assessment will be administered to participants immediately after intervention.
  The Montreal Cognitive Assessment is a cognitive screening assessment that is used to measure several cognitive domains, which include working memory, delayed recall, visuospatial abilities, executive functions, attention, concentration, language, and orientation to time and place. The total score ranges from 0 to 30. One extra point is added to adjust the total score for participants who received less than 12 years of education.
The Chedoke Arm and Hand Activity Inventory | The Chedoke Arm and Hand Activity Inventory will be administered to participants at baseline.
  The CAHAI evaluates the functional ability of the affected arm and hand to perform tasks after stroke. The 13 items contained in the CAHAI represent bimanual meaningful everyday activities and are made up a variety of the upper-extremity characteristics, including strength, dexterity, coordination, and grasp. The 7-point activity scale is used in the CAHAI, where 1 indicates "performing less than 25% of the effort to complete the task" and 7 indicates "the participants' affected upper extremity is able to complete the task competently independently." The reliability and validity of the CAHAI have been ascertained in stroke.
The Chedoke Arm and Hand Activity Inventory | The Chedoke Arm and Hand Activity Inventory will be administered to participants immediately after intervention.
  The CAHAI evaluates the functional ability of the affected arm and hand to perform tasks after stroke. The 13 items contained in the CAHAI represent bimanual meaningful everyday activities and are made up a variety of the upper-extremity characteristics, including strength, dexterity, coordination, and grasp. The 7-point activity scale is used in the CAHAI, where 1 indicates "performing less than 25% of the effort to complete the task" and 7 indicates "the participants' affected upper extremity is able to complete the task competently independently." The reliability and validity of the CAHAI have been ascertained in stroke.
The Chedoke Arm and Hand Activity Inventory | The Chedoke Arm and Hand Activity Inventory will be administered to participants three months after intervention.
  The CAHAI evaluates the functional ability of the affected arm and hand to perform tasks after stroke. The 13 items contained in the CAHAI represent bimanual meaningful everyday activities and are made up a variety of the upper-extremity characteristics, including strength, dexterity, coordination, and grasp. The 7-point activity scale is used in the CAHAI, where 1 indicates "performing less than 25% of the effort to complete the task" and 7 indicates "the participants' affected upper extremity is able to complete the task competently independently." The reliability and validity of the CAHAI have been ascertained in stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Keh-chung Lin, ScD, Principal Investigator — National Taiwan University
Locations (2):
- Taiwan (2):
  - Fongyuan Hospital, Taichung
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YC, Li YC, Lin KC, Chen CL, Wu YH, Kuo C, Yeh YP, Liu TX. Effects of proximal priority and distal priority robotic priming techniques with impairment-oriented training of upper limb functions in patients with chronic stroke: study protocol for a single-blind, randomized controlled trial. Trials. 2021 Sep 8;22(1):604. doi: 10.1186/s13063-021-05561-6. PMID 34496938